CLINICAL TRIAL: NCT00622323
Title: Post Marketing Surveillance Study of Byetta ™ (Exenatide) Use Among Filipino Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: H8O-PH-B006; H8O-PH-B006
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; metformin; sulfonylurea; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-interventional, post marketing surveillance study to determine the proportion of patients experiencing an adverse event and a list of the experienced adverse events, serious and non-serious, that would occur among Filipino patients with type 2 diabetes mellitus who are treated with exenatide who are taking metformin, a sulfonylurea or a combination of metformin and a sulfonylurea but have not achieved adequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* are male or female outpatients at least 18 years of age
* provide written consent to the release of their data after being informed of the study
* diagnosed with type 2 diabetes mellitus and are taking metformin, or a sulfonylurea or both
* are reliable, and agree to keep all appointments for clinic visits, complete tests and procedures as may be required by the attending physician in the course of routine clinical care
* are treated with exenatide according to the approved Product Insert, as prescribed by the investigator in the routine care of the patient

Exclusion Criteria:

* are simultaneously participating in a different study that includes a treatment intervention and/or an investigational drug.
* are currently taking insulin.
* are pregnant or have intentions of becoming pregnant within the duration of the study.
* are the investigators or their immediate families. Immediate family is defined as the investigator's spouse, parents, natural or legally adopted child (including stepchild living in the investigator's household), grandparents, or grandchild. Employees of investigators are also not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients at least 18 years of age and diagnosed with type 2 diabetes mellitus treated in an ambulatory care setting and who are taking metformin, a sulfonylurea, or a combination of metformin and sulfonylurea, but have not achieved adequate glycemic control. Female patients eligible of becoming pregnant are required to have some form of contraception while participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients experiencing an adverse event and a list of the experienced adverse events, that would occur among Filipino patients with type 2 diabetes and inadequate glycemic control treated with exenatide | 12 weeks

SECONDARY OUTCOMES:
To evaluate the change from baseline to endpoint in HbA1c and body weight of Filipino patients with type 2 diabetes mellitus treated with exenatide who are taking metformin and/or a sulfonylurea but have not achieved adequate glycemic control. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (3):
- Philippines (3):
  - Research Site, Paranaque City
  - Research Site, Pasig
  - Research Site, Taytay

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com/